CLINICAL TRIAL: NCT06780605
Title: Observational Study to Investigate the Correlation of the Genetic Constitution of the Spent Blastocyst Media (SBM) With the Inner Cell Mass (ICM) and Multifocal Trophectoderm (TE) Biopsies
Brief Title: Correlation of the Genetic Constitution of the Spent Blastocyst Media
Acronym: CONNECTED
Status: Completed | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX1-GCO-CR-23-04
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Infertility (IVF Patients)
Keywords: PGT-A; Trophectoderm; Inner cell mass; Blastocyst; Infertility; In vitro fertilization; niPGT-A; Embryo development; Embryonic cell-free DNA; Embryo selection
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies of blastocyst trophectoderm and inner cell mass. Spent blastocyst media with embryonic cell-free DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Embryos donated for research after an assisted reproduction treatment: Study specific procedures will start only when the potential participant couples have undergone their scheduled IVF/ICSI and/or PGT-A cycles following clinics´ standard practice to obtain blastocysts that will be vitrified. If they accept to donate the surplus blastocysts not used in their reproductive treatment to the current study by signing the informed consent, lab operators will carry out embryo warming and will select the appropriate blastocysts to go through the study protocol procedures (collection of SBM and TE/ICM biopsies). No drugs or medical devices will be used.
  Interventions: Genetic: niPGT-A; Genetic: Multifocal TE biopsies and ICM biopsy

INTERVENTIONS:
Genetic: niPGT-A — After being thawed following the standard lab practice, any donated blastocyst usable for the study will be washed individually to remove any trace of cumulus DNA and will be transferred to a new culture dish with a drop of 10-15µl. Day-5 blastocysts with proper re-expansion after thawing, will be cultured overnight (≈24 hours) before media collection and TE/ICM biopsies. Day-6 blastocysts will be cultured a total of 8 hours after thawing, before media collection and TE/ICM biopsies.
  On day 6/7, the embryos' media will be collected with an automatic pipette for niPGT-A and additional genetic analysis. The same protocol will be used to analyze SBM and blastocyst biopsies.
Genetic: Multifocal TE biopsies and ICM biopsy — For biopsy, blastocysts will be transferred to the biopsy dish and multi-focal TE biopsies will be performed in three locations related to the position of the ICM. ICM biopsies will be performed following a published protocol provided to the participant centers. ICM and TE sections will be aspirated with the use of micropipettes adapted to a micromanipulation and laser microscope system.
  For the genetic study of the samples, the same protocol will be used to analyze embryo biopsies and SBM.

SUMMARY:
The main objective of this study is to improve niPGT-A (non-invasive Preimplantation Genetic Testing for Aneuploidies) to avoid the need of a biopsy to perform the genetic analysis of the embryo and to help in understanding the genetic constitution of different parts of the blastocyst (early stage of an embryo development).

For this purpose, we aim to analyses the genetic material released by the embryo to the culture medium (also called Spent Blastocyst Media, SBM) from about 200 blastocysts donated to research by participants of assisted reproduction treatments.

The results will be correlated with the ones obtained from performing the same analysis on biopsies taken from the outer (trophectoderm, TE) and the inner (inner cell mass, ICM) layer of cells in different locations to investigate the mechanisms and origin of the blastocyst genetic content released to the culture medium during preimplantation embryo development.

DETAILED DESCRIPTION:
The study and selection of embryos before transfer is a key step for the success of infertility treatments in assisted reproduction. The current techniques applied are called preimplantation genetic testing of aneuploidies (PGT-A) and are highly sensitive and specific, although they require the retrieval of four to six cells (a biopsy) from an embryo at an early stage of development (blastocyst stage).

Nowadays, the alternatives for embryo selection given to young and healthy women or to couples that do not want to undergo PGT-A are based on studying the morphology and development of the embryos. Unfortunately, these are not reliable methods to know if the embryos have the right number of chromosomes.

A new method called non-invasive PGT-A (niPGT-A) analyses the genetic material released by the embryo to the culture medium (Spent Blastocyst Media, SBM) where the embryo grows in the IVF lab. This genetic material allows for identification of the chromosome number of the embryo. In a previous pilot study, the results of the analysis of the culture media were concordant with the results of the embryo biopsy in 85% of cases.

The current study will analyze the genetic constitution of the SBM and correlate the results of the same analysis on the inner cell mass (ICM) and trophectoderm (TE) cells taken in different locations (multifocal biopsy) to improve our understanding of the mechanisms and origin of the embryo genetic content released to the culture medium during its preimplantational development.

Once this prospective and observational study is approved by the competent Research Ethics Committee, the recruitment and selection of patients will follow. Every potential participant will be asked to sign the study informed consent only after finishing their assisted reproductive treatment.

To comply with the design of this pilot study, a total number of 200 blastocysts donated to research after IVF/ICSI or PGT-A cycles has been estimated to generate enough results. After warming, blastocysts will be subjected to multifocal biopsies of TE, ICM isolation and collection of the SBM. This part of the study will be performed in the collaborating centers. Samples will be shipped to Igenomix Spain for the genetic research and further data analysis.

The expected duration of the study is 18 months. Embryos will be included in the different participating centers for an estimated period of 9 months. Participants involvement in the study is just linked to the moment of the consent form signature for the embryo donation. This study will not imply any modification of a scheduled IVF/ICSI or PGT-A cycles nor extra visits to the recruiting centers.

ELIGIBILITY:
Inclusion Criteria:

* Study informed consent form, approved by the Ethics Committee, signed.
* Any patient with aneuploid or euploid blastocysts from PGT-A cycles donated for research.
* Patients undergoing regular IVF/ICSI cycles aiming to donate surplus embryos for research.
* Embryos from own or donated oocytes can be included.
* Embryos fertilized with donated sperm can be included.
* Only blastocysts with proper re-expansion and good quality after thawing will be included.

Exclusion Criteria:

* Blastocysts that had not survived to vitrification, that had not re-expanded properly or having poor ICM or TE quality.

Note: No exclusion criteria specific to the patients' background will be considered.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Donated embryos to research from patients undergoing IVF/ICSI or PGT-A cycles will be eligible for the study after informed consent signature.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Chromosomal status of the embryos | Up to 6/7 days of embryo development
  Concordance of the genetics results between SBM and TE and ICM biopsies samples analysis results.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Mir Pardo, PhD, Principal Investigator — Igenomix; Luis Navarro Sanchez, PhD, Principal Investigator — Igenomix
Locations (2):
- Cyprus (2):
  - British Cyprus IVF Hospital, Nicosia
  - Ventus IVF Center, Nicosia

IPD SHARING:
Plan to Share IPD: No